CLINICAL TRIAL: NCT05346328
Title: An Open-clinical Trial Phase Ⅱ, Injection of A166 for HER2-positive Patients With Refractory Unresectable Locally Advanced or Metastatic Breast Cancer；KL166-IIS-001
Brief Title: HER2-positive Breast Cancer Project Initiated by Investigators
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Fudan University (Other)
Responsible Party: Principal Investigator, Xichun Hu, Chief Physician, Fudan University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: KL166-IIS-001
Record Dates: First submitted 2022-01-14; First posted 2022-04-26 (Actual); Last update posted 2022-04-26 (Actual); Status verified 2022-04

CONDITIONS: Breast Cancer
Keywords: HER2-positive Breast Cancer
MeSH Terms: conditions — Breast Neoplasms

STUDY DESIGN:
Intervention Model Description: This study adopts an open research design and selects patients with refractory HER2-positive unresectable locally advanced or metastatic breast cancer who have failed previous ADC drug treatment. The patients who met the enrollment conditions were treated with injection of A166.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Single Group Assignment (Experimental): This study adopts an open research design and selects patients with refractory HER2-positive unresectable locally advanced or metastatic breast cancer who have failed previous ADC drug treatment. The patients who met the enrollment conditions were treated with injection of A166.
  Interventions: Drug: Injection of A166

INTERVENTIONS:
Drug: Injection of A166 — 4.8 mg/kg for each 21 (±3) -day cycle

SUMMARY:
This study will assess the objective response rate (ORR), safety, progression-free survival (PFS) , overall survival (OS), 6-month survival rate, 12-month survival rate, 18-month survival rate, 24-month survival rate, disease control rate (DCR), clinical benefit rate (CBR), duration of response (DOR) and Time to Response (TTR). Injection of A166 for HER2-positive patients with refractory unresectable locally advanced or metastatic breast cancer who have failed previous ADC drug therapy.

ELIGIBILITY:
Inclusion Criteria:

* 1. Male or female patient ≥ 18 years and ≤ 75 years when signing the informed consent form; 2. Breast cancer patients by histopathology and/or cytology documented, including:

  a) Participants with unresectable locally advanced or metastatic breast cancer; b) Evaluated or tested as HER2-positive expression. The definition of HER2 positive in this study: immunohistochemistry (IHC) was 2+ and confirmed by fluorescence in situ hybridization (FISH), or IHC was 3+; 3. Have received at least 3 targeted therapies for locally advanced or metastatic disease, including:
  1. Disease progression after receiving at least 1 trastuzumab-containing (including a biosimilar of trastuzumab on the market)-based treatment;
  2. After receiving at least one anti-HER2 tyrosine kinase inhibitor (lapatinib or pyrrotinib)-based treatment plan, the disease progresses or cannot tolerate toxic and side effects;
  3. The disease progresses or cannot tolerate toxic and side effects after receiving treatment with antibody-conjugated drugs targeting HER2 (such as T-DM1 or other ADCs); Note: Adjuvant therapy and anti-HER2 therapy used in the neoadjuvant treatment stage before radical treatment are not counted, but recurrence or metastasis occurs during the last anti-HER2 medication period or within one year after the end, it can be regarded as a plan.

     4. Have previously received taxanes to treat breast cancer;

     Exclusion Criteria:
* 1. Serious or uncontrollable heart diseases that require treatment, including:

  1. Congestive heart failure graded 3 or 4 by the New York College of Cardiology (NYHA);
  2. Unstable angina pectoris that cannot be controlled by drugs;
  3. Myocardial infarction occurred within 6 months before the first administration of the study treatment;
  4. Severe arrhythmia requiring medical treatment (except for atrial fibrillation or paroxysmal supraventricular tachycardia); 2. Baseline measurement, QTc interval, male> 450 msec, female> 470 msec; 3. Clinically active interstitial lung disease; 4. Patients with primary central nervous system (CNS) malignant tumors or CNS metastases that have failed local treatment; for asymptomatic brain metastases, or with stable clinical symptoms and no need for steroids and other brain metastases within 4 weeks before the first administration of the trial drug Treated patients can be included in the group; 5. Those who are known to have a history of hypersensitivity to other monoclonal antibodies or allergic to A166 and its components for injection; 6. Those who have permanently discontinued trastuzumab due to any toxicity;

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 48 (Estimated)
Dates: Start 2022-06-01 (Estimated); Primary Completion 2023-12-31 (Estimated); Study Completion 2024-12-31 (Estimated)

PRIMARY OUTCOMES:
Objective response rate（ORR） | 2 years
  ORR is defined as the percentage of subjects who have achieved complete response and partial response according RECIST 1.1.

SECONDARY OUTCOMES:
Progression-free survival(PFS) | 2 years
  PFS is defined as the time between date of first dose of study therapy and date of progression or death according RECIST 1.1.
Disease control rate(DCR) | 2 years
  DCR is defined as cases where objective remission(assessed as complete remission or partial remission according RECIST 1.1 standard) or stable disease during the study.
Clinical benefit rate(CBR) | 2 years
  CBR is defined as the proportion of patients with a complete or partial response or with stable disease according RECIST 1.1
Duration of rate(DOR) | 2 years
  DOR is defined the time between the first tumor evaluation for CR or PR and the first evaluation for PD(Progressive Disease) or death from any cause according RECIST 1.1.
Time to response(TTR) | 2 years
  TTP is defined as the time between randomization and objective tumor progression according RECIST 1.1; TTP does not include death
Overall survival(OS) | 2 years
  Overall survival(OS) is defined as the time from first dose of study therapy to the date of death(any case).Subjects who are alive censored at the last known time that the subject was alive.

CONTACTS AND LOCATIONS:
Overall Officials: Xichun Hu, Doctor, Principal Investigator — Chief Physician

REFERENCES:
- [Result] Krop IE, Kim SB, Gonzalez-Martin A, LoRusso PM, Ferrero JM, Smitt M, Yu R, Leung AC, Wildiers H; TH3RESA study collaborators. Trastuzumab emtansine versus treatment of physician's choice for pretreated HER2-positive advanced breast cancer (TH3RESA): a randomised, open-label, phase 3 trial. Lancet Oncol. 2014 Jun;15(7):689-99. doi: 10.1016/S1470-2045(14)70178-0. Epub 2014 May 2. PMID 24793816
- [Result] Krop IE, Kim SB, Martin AG, LoRusso PM, Ferrero JM, Badovinac-Crnjevic T, Hoersch S, Smitt M, Wildiers H. Trastuzumab emtansine versus treatment of physician's choice in patients with previously treated HER2-positive metastatic breast cancer (TH3RESA): final overall survival results from a randomised open-label phase 3 trial. Lancet Oncol. 2017 Jun;18(6):743-754. doi: 10.1016/S1470-2045(17)30313-3. Epub 2017 May 16. PMID 28526538
- See also: Related Info — http://pubmed.ncbi.nlm.nih.gov/24793816/
- See also: Related Info — http://pubmed.ncbi.nlm.nih.gov/28526538/